CLINICAL TRIAL: NCT00879437
Title: A Phase 2 Study of Valproic Acid and Radiation, Followed by Maintenance Valproic Acid and Bevacizumab in Children With Newly Diagnosed High-grade Gliomas or Brainstem Gliomas
Brief Title: Valproic Acid, Radiation, and Bevacizumab in Children With High Grade Gliomas or Diffuse Intrinsic Pontine Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Cook Children's Medical Center (Other); University of Oklahoma (Other); University of Texas, Southwestern Medical Center at Dallas (Other); The University of Texas Health Science Center at San Antonio (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Jack Su, MD, Study Chair, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24549
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Glial Cell Tumors; Malignant Gliomas; Glioblastoma Multiforme; Anaplastic Astrocytoma; Gliomatosis Cerebri; Gliosarcoma; Brainstem Glioma; Diffuse Intrinsic Pontine Glioma
Keywords: brain tumor; bevacizumab; valproic acid; radiation therapy
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Neoplasms, Neuroepithelial; Gliosarcoma; Diffuse Intrinsic Pontine Glioma; Brain Neoplasms | interventions — Valproic Acid; Bevacizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- valproic acid and radiation, followed by valproic acid and bevacizumab (Experimental): radiation phase (week 1-6): daily valproic acid and radiation, for approximately 6 weeks post-radiation phase (week 7-10): valproic acid daily maintenance phase (starting week 11): daily valproic acid, and bevacizumab once every 2 weeks; to continue for a maximum duration of 2 years
  Interventions: Drug: Valproic acid; Drug: Bevacizumab; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Valproic acid — Daily (pre-XRT, During XRT, Post-XRT and Maintenance Therapy) Started at 15 mg/kg/day divided into three doses a day as soon as patients have recovered from surgery but no later than the first day of XRT.
  Dosage will be adjusted in increments of 5 mg/kg/day every 3-5 days to achieve and maintain trough concentrations between 85 and 115 mcg/ml
  Other Names: sodium valproate
Drug: Bevacizumab — All patients will receive bevacizumab (10 mg/kg iv) during the maintenance phase every two weeks for a maximum duration of therapy of 24 months.
  Other Names: Avastin
Radiation: Radiation therapy — Radiation therapy will start within 30 days of the definitive surgical procedure. Primary brain malignant gliomas will receive a total dose of between 54.0 and 59.4 Gy in 30-33 fractions over 6-7 weeks. Total dose will be 54.0 Gy for completely resected tumors and brainstem gliomas. The total dose will be 59.4 if the tumor is located in the brain but not the brainstem, and the tumor was incompletely resected. Primary spinal cord malignant gliomas will receive a total dose of between 50.4-54 Gy in 28-30 fractions over 5-6 weeks.

SUMMARY:
Currently, there are few effective treatments for the following aggressive brain tumors: glioblastoma multiforme, anaplastic astrocytoma, gliomatosis cerebri, gliosarcoma, or brainstem glioma. Surgery and radiation can generally slow down these aggressive brain tumors, but in the majority of patients, these tumors will start growing again in 6-12 months. Adding chemotherapy drugs to surgery and radiation does not clearly improve the cure rate of children with malignant gliomas.

The investigators are conducting this study to see if the combination of valproic acid and bevacizumab (also known as AvastinTM) with surgery and radiation will shrink these brain tumors more effectively and improve the chance of cure.

DETAILED DESCRIPTION:
With the exception of patients with diffuse intrinsic pontine glioma (DIPG), all patients should have the maximal surgical resection that can be safely performed prior to study entry. Submission of frozen tumor is strongly encouraged. After recovery from neurosurgery, all patients will start valproic acid (VPA) and radiation therapy.

VPA will be started at 15 mg/kg/day divided into three doses a day, ideally 48 hours prior to first day of radiation therapy, but no later than the first day of radiation therapy. Patients may also begin VPA sooner if they have post-operative seizures and require an anti-convulsant.

Radiation phase (week 1-6): Radiation therapy should begin within 30 days of definitive surgery or radiographic diagnosis, whichever is the later date. Date of surgery or radiographic diagnosis is considered day 1, and radiation should start no later than day 31. VPA will be continued daily without interruption during radiation therapy. VPA doses will be adjusted in increments of 5 mg/kg/day every 3-5 days to achieve and maintain trough concentrations between 85 to 115 mcg/ml. All patients will receive standard radiation therapy which will last approximately six week.

Post Radiation Phase (week 7-10): Patients will continue to receive VPA as previously dosed during radiation to maintain a trough concentration of 85-115 mcg/ml.

Maintenance Phase (starting week 11): Maintenance therapy will begin approximately 4 weeks after completion of radiation or week 11, whichever comes first.

Patients will continue VPA daily during maintenance therapy. All patients will start bevacizumab, 10 mg/kg intravenously every two weeks, at the start of maintenance therapy (week 11). Maintenance therapy will continue uninterrupted unless treatment related toxicities requires study drug interruption. In the absence of unacceptable toxicity or disease progression, patients will continue to receive protocol treatment for a maximum duration of two years (including the radiation phase).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be greater than or equal to 3 years and less than or equal to 21 years of age at the time of study enrollment.
2. Patients must have histologic verifications of a glioblastoma multiforme, anaplastic astrocytoma, gliomatosis cerebri (WHO grade III or IV glioma with diffuse parenchymal and/or leptomeningeal involvement), or gliosarcoma at the time of study enrollment. Patients with newly diagnosed intrinsic brainstem gliomas, defined as tumors with a pontine epicenter and diffuse rather than focal involvement of th pons, with or without extension to adjacent medulla or midbrain, are eligible without histologic confirmation. Patients with brainstem tumors that do not meet these criteria or not considered to be typical intrinsic pontine gliomas will only be eligible if the tumors are biopsied and proven to be a grade III or IV glioma (anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma).
3. Patients must have Karnofsky Performance Score (for patients greater than 16 years of age) or Lansky Performance Score (for patients less than or equal to 16 years of age) greater than or equal to 50% assessed within two weeks of study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
4. Patients must not have received any prior chemotherapy, radiation therapy, biologic therapy, or bone marrow transplant. Surgery and dexamethasone are permitted prior to study entry. In patients who require anti-convulsant prior to study entry, it is permissible to start VPA, but trough VPA concentration must be repeated within 48 hours of study entry.
5. Patients must have adequate bone marrow function defined as: - Hgb greater than or equal to 8 gm/dL (transfusion independent) - Platelet count greater than or equal to 100,000/mm3 (transfusion independent) - Absolute neutrophil count (ANC) greater than or equal to 1,000/ mm3
6. Patients must have adequate liver function defined as:

   * Bilirubin (sum of conjugated + unconjugated) less than or equal to 1.5 times institutional upper limit of normal (ULN) for age.
   * SGPT (ALT) less than or equal to 2.5 times institutional ULN for age.
   * Serum albumin greater than or equal to 2 g/dL.
7. Patients must have adequate renal function defined as:

   * Urine protein (albumin)/creatinine ratio of less than 1.0
   * Creatinine clearance or radioisotope GFR greater than or equal to 70 ml/min/1.73m2 OR
   * A serum creatinine based on age and gender as follows:

     * 2 to less than 6 years of age: 0.8 mg/dL for male and female
     * 6 to less than 10 year of age: 1.0 mg/dL for male and female
     * 10 to less than 13 years of age: 1.2 mg/dL for male and female
     * 13 to less than 16 years of age: 1.5 mg/dL for males and 1.4 for females
     * Greater than or equal to 16 years of age: 1.7 mg/dL for males and 1.4 mg/dL for females

   Note: The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.
8. Amylase and lipase less than or equal to 2 times institutional ULN for age.
9. Patients must not have a prolonged PT or PTT (greater than 1.2 times the institutional upper limit of normal), and the INR must be less than 1.5.
10. MRI ECHO gradient sequences are required to evaluate for the presence or absence of CNS hemorrhage. Patients with intra-tumoral and/or CNS hemorrhage are eligible for study entry if they fulfill the following guidelines:

    * Patients with an asymptomatic intra-tumoral/intracranial hemorrhage measuring less than 1 cm in the widest dimension on MRI at the time of diagnosis, after surgery, and/or any time prior to study enrollment, are eligible; hemorrhage must not have progressed on MRI prior to initiation of protocol therapy; patients mut not have developed progressive symptoms thought to be related to the intra-tumoral/intracranial hemorrhage prior to initiation of protocol therapy.
    * Patients with a greater than 1 asymptomatic intra-tumoral/intracranial hemorrhage but all measuring less than 1 cm in the widest dimension on MRI are eligible if they fulfill the guidelines described above.
    * Patients with asymptomatic post-operative hemorrhage in and/or around the surgical cavity are eligible for study entry if they otherwise fulfill the guidelines described above.
    * Patients with an intra-tumoral hemorrhage greater than 1 cm at diagnosis but who demonstrate minimal post-operative hemorrhage as described above after tumor resection are eligible for study.
11. Patients must begin radiation therapy within 30 days of surgery or radiographic diagnosis, whichever is the later date.
12. All patients and/or their legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

1. Females of reproductive potential must not be pregnant or lactating. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
2. Patients with active or history of cardiac (CHF, myocardial infarction, myocarditis) disease are excluded from this trial.
3. Patients receiving any of the following medications are not eligible for study entry: a. Anti-cancer therapy or investigational agents b.Anti-coagulants (except for heparin to maintain the patency of central venous catheters). c.Growth factors for white blood cell, red blood cell or platelet support d.Aspirin (> 81 mg/day) e.Non-steroidal anti-inflammatory drugs f.Clopidogrel (Plavix), Dypiramidole (Persantine), or any other drug that inhibits platelet function g. Anti-convulsants: patients on any anti-convulsant with the exception of VPA are eligible for study entry. It is strongly recommended that a neurology consult be obtained to enable discontinuation of all anti-convulsant other than VPA, whenever possible.
4. Patients who have an uncontrolled infection are not eligible.
5. Patients with inadequately controlled systemic hypertension (SBP and/or DBP greater than 95th percentile for age and height)
6. Patients with a prior history of hypertensive crisis and/or hypertensive encephalopathy

   If a BP measurement prior to registration is greater than 95th percentile for age and height, it must be rechecked and documented to be less than 95th percentile for age and height prior to registration. If a patient falls between the height or weight percentiles, site should average the value as appropriate. For patients greater than or equal to 18 years, use adult normal ranges for blood pressure. Patients with hypertension are eligible if their blood pressures become less than 95th percentile after anti hypertensive medications.
7. Prior Ischemic Events: Patients with a history of stroke, myocardial infarction, or unstable angina within 6 months prior to registration are not eligible.
8. Vascular Disease: Patients with significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to registration will not be eligible.
9. Patients with a history of hemoptysis, bleeding diathesis, known platelet disorder, or coagulopathy are not eligible.
10. Patients with a history of abdominal fistula or GI perforation within 6 months prior to registration are not eligible.
11. Patients with a known or suspected urea cycle or other metabolic disorder are not eligible.
12. Patients with abnormality of the tibial metaphyseal plate on plain X-ray prior to study entry are not eligible.
13. Patients with a history of a serious non-healing wound, ulcer, or bone fracture are not eligible.
14. Patients with any clinically significant systemic illness, including serious infection, pulmonary, hepatic, or other organ impairment, that would compromise tolerance and/or timely completion of protocol therapy.

16. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements and/or follow-up studies of this trial.

17. Patients with a known hypersensitivity to any component of bevacizumab are not eligible for this trial.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2015-08-30 (Actual); Study Completion 2017-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Su, MD, Study Chair — Baylor College of Medicine
Locations (6):
- United States (6):
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Medical Center Dallas, Center for Cancer and Blood Disorders, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Results of this study has been published (Su JM, et al., Pediatr Blood Cancer 2020: 67:e28283). Additional de-identified information can be provided upon request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Results of this study has been published (Su JM, et al., Pediatr Blood Cancer 2020: 67:e28283). Additional de-identified information can be provided upon request.
Access Criteria: Pediatr Blodd Cancer 2020 Jun;67(6):e28283. doi: 10.1002/pbc.28283. PMID: 32285998.
URL: https://pubmed.ncbi.nlm.nih.gov/32285998/

REFERENCES:
- [Result] Su JM, Murray JC, McNall-Knapp RY, Bowers DC, Shah S, Adesina AM, Paulino AC, Jo E, Mo Q, Baxter PA, Blaney SM. A phase 2 study of valproic acid and radiation, followed by maintenance valproic acid and bevacizumab in children with newly diagnosed diffuse intrinsic pontine glioma or high-grade glioma. Pediatr Blood Cancer. 2020 Jun;67(6):e28283. doi: 10.1002/pbc.28283. Epub 2020 Apr 14. PMID 32285998
- See also: Results of this trial has been peer-reviewed and published — https://pubmed.ncbi.nlm.nih.gov/32285998/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled between September 2009 through August 2015, from five participating sites.
Pre-assignment Details: A total of 38 eligible patients, 20 diffuse intrinsic pontine glioma (DIPG), and 18 high-grade glioma (HGG), were enrolled from five institutions.
Groups:
- Diffuse Intrinsic Pontine Gliomas (DIPG): Newly diagnosed diffuse intrinsic pontine gliomas; a total of 20 patients enrolled
  treatment description: radiation phase (week 1-6): daily valproic acid and radiation, for approximately 6 weeks post-radiation phase (week 7-10): valproic acid daily maintenance phase (starting week 11): daily valproic acid, and bevacizumab once every 2 weeks; to continue for a maximum duration of 2 years
  Valproic acid: Daily (pre-XRT, During XRT, Post-XRT and Maintenance Therapy) Started at 15 mg/kg/day divided into three doses a day as soon as patients have recovered from surgery but no later than the first day of XRT.
  Dosage will be adjusted in increments of 5 mg/kg/day every 3-5 days to achieve and maintain trough concentrations between 85 and 115 mcg/ml
  Bevacizumab: All patients will receive bevacizumab (10 mg/kg iv) during the maintenance phase every two weeks for a maximum duration of therapy of 24 months.
  Radiation therapy: Radiation therapy will start within 30 days of the definitive surgical procedure. Primary brain malignant gliomas will receive a total dose of between 54.0 and 59.4 Gy in 30-33 fractions over 6-7 weeks. Total dose will be 54.0 Gy for completely resected tumors and brainstem gliomas. The total dose will be 59.4 if the tumor is located in the brain but not the brainstem, and the tumor was incompletely resected. Primary spinal cord malignant gliomas will receive a total dose of between 50.4-54 Gy in 28-30 fractions over 5-6 weeks.
- High-grade Gliomas (HGG): Newly diagnosed high grade gliomas; a total of 18 patients enrolled
  treatment description: radiation phase (week 1-6): daily valproic acid and radiation, for approximately 6 weeks post-radiation phase (week 7-10): valproic acid daily maintenance phase (starting week 11): daily valproic acid, and bevacizumab once every 2 weeks; to continue for a maximum duration of 2 years
  Valproic acid: Daily (pre-XRT, During XRT, Post-XRT and Maintenance Therapy) Started at 15 mg/kg/day divided into three doses a day as soon as patients have recovered from surgery but no later than the first day of XRT.
  Dosage will be adjusted in increments of 5 mg/kg/day every 3-5 days to achieve and maintain trough concentrations between 85 and 115 mcg/ml
  Bevacizumab: All patients will receive bevacizumab (10 mg/kg iv) during the maintenance phase every two weeks for a maximum duration of therapy of 24 months.
  Radiation therapy: Radiation therapy will start within 30 days of the definitive surgical procedure. Primary brain malignant gliomas will receive a total dose of between 54.0 and 59.4 Gy in 30-33 fractions over 6-7 weeks. Total dose will be 54.0 Gy for completely resected tumors and brainstem gliomas. The total dose will be 59.4 if the tumor is located in the brain but not the brainstem, and the tumor was incompletely resected. Primary spinal cord malignant gliomas will receive a total dose of between 50.4-54 Gy in 28-30 fractions over 5-6 weeks.
Period: Overall Study
Arm/Group | Diffuse Intrinsic Pontine Gliomas (DIPG) | High-grade Gliomas (HGG)
Started | 20 | 18
Completed | 19 | 17
Not Completed | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: 20 participants with diffuse intrinsic pontine gliomas; 18 patients with high-grade gliomas
Groups:
- Valproic Acid and Radiation, Followed by Valproic Acid and Bevacizumab: radiation phase (week 1-6): daily valproic acid and radiation, for approximately 6 weeks post-radiation phase (week 7-10): valproic acid daily maintenance phase (starting week 11): daily valproic acid, and bevacizumab once every 2 weeks; to continue for a maximum duration of 2 years
  Valproic acid: Daily (pre-XRT, During XRT, Post-XRT and Maintenance Therapy) Started at 15 mg/kg/day divided into three doses a day as soon as patients have recovered from surgery but no later than the first day of XRT.
  Dosage will be adjusted in increments of 5 mg/kg/day every 3-5 days to achieve and maintain trough concentrations between 85 and 115 mcg/ml
  Bevacizumab: All patients will receive bevacizumab (10 mg/kg iv) during the maintenance phase every two weeks for a maximum duration of therapy of 24 months.
  Radiation therapy: Radiation therapy will start within 30 days of the definitive surgical procedure. Primary brain malignant gliomas will receive a total dose of between 54.0 and 59.4 Gy in 30-33 fractions over 6-7 weeks. Total dose will be 54.0 Gy for completely resected tumors and brainstem gliomas. The total dose will be 59.4 if the tumor is located in the brain but not the brainstem, and the tumor was incompletely resected. Primary spinal cord malignant gliomas will receive a total dose of between 50.4-54 Gy in 28-30 fractions over 5-6 weeks.
Arm/Group | Valproic Acid and Radiation, Followed by Valproic Acid and Bevacizumab
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 29
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: 1-year Event Free Survival (EFS)
Description: To compare 1-year EFS for this trial versus historical series (ACNS0126 for high-grade gliomas; CCG-9941 for DIPG)
Time Frame: 12 months
Population: 1 patient with DIPG not evaluable due to early death (did not complete valproic acid and radiation) related to a surgical complication (unrelated to protocol therapy)
  1 patient with HGG not evaluable due to non-compliance with protocol therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Diffuse Intrinsic Pontine Glioma: 20 eligible patients, 19 evaluable patients
- High-grade Gliomas: 18 eligible patients, 17 evaluable patients
Arm/Group | Diffuse Intrinsic Pontine Glioma | High-grade Gliomas
Number analyzed (Participants) | 19 | 17
percentage of participants | 12 [2 to 31] | 24 [7 to 45]
Statistical Analysis 1: Comparison: Diffuse Intrinsic Pontine Glioma vs High-grade Gliomas; comparing 1-year EFS of DIPG on this trial versus historical control (1-year EFS of 17% from CCG-9941; PMID 12177103) comparing 1-year EFS of HGG on this trial versus historical control (1-year EFS of 36% from ACNS0126; PMID 21339192); Test type: Non-Inferiority — if 19 evaluable patients enrolled for DIPG, study is powered at 80% to detect a 20% improvement in 1-year EFS compared to historical control if 21 evaluable patients enrolled for HGG, study is powered at 80% to detect a 20% improvement in 1-year EFS compared to historical control; p < 0.05, Log Rank; one sample log-rank

2. Primary Outcome: Percentage of Participants With Grade 3 Thrombocytopenia Assessed by CTCAE v3.0 During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 3 thrombocytopenia, graded according to CTCAE v3.0, during concurrent valproic acid and radiation treatment for week 1-10
Time Frame: first 10 weeks of study
Measure: Count of Participants; unit: Participants
Groups:
- 38 Eligible Patients: 38 eligible patients, regardless of tumor type
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

3. Primary Outcome: Percentage of Participants With Grade 3 Neutropenia Assessed by CTCAE v3.0 During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 3 neutropenia, graded by CTCAE v3.0, during concurrent valproic acid and radiation treatment for the first 10 weeks
Time Frame: first 10 weeks of study
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 3

4. Primary Outcome: Percentage of Participants With Grade 3 Lymphopenia Assessed by CTCAE v3.0 During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 3 lymphopenia, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of study
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 5

5. Primary Outcome: Percentage of Participants With Grade 3 Leukopenia, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 3 leukopenia, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of study
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

6. Primary Outcome: Percentage of Participants With Grade 2 Somnolence, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 2 somnolence, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of study
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

7. Primary Outcome: Percentage of Participants With Grade 2 Fatigue, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 2 fatigue, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of study
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 3

8. Primary Outcome: Percentage of Participants With Grade 3 Weight Gain, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 3 weight gain, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment during week 1-10
Time Frame: first 10 weeks of study
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

9. Primary Outcome: Percentage of Participants With Grade 2 Weight Gain, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 2 weight gain, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of study
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 4

10. Primary Outcome: Percentage of Participants With Grade 2 Hypoglycemia, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 2 hypoglycemia, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of study
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

11. Primary Outcome: Percentage of Participants With Grade 3 Lipase and Amylase Elevation, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 3 lipase and amylase elevation, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

12. Primary Outcome: Percentage of Participants With Grade 2 Pancreatitis, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 2 pancreatitis, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of study
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

13. Primary Outcome: Percentage of Participants With Grade 3 Dehydration, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 3 dehydration, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

14. Primary Outcome: Percentage of Participants With Grade 4 Radiation Necrosis, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 4 radiation necrosis, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

15. Primary Outcome: Percentage of Participants With Grade 2 Abdominal Pain, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 2 abdominal pain, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment, week 1-10
Time Frame: first 10 weeks of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

16. Primary Outcome: Percentage of Participants With Grade 2 AST Elevation, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 2 AST elevation, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

17. Primary Outcome: Percentage of Participants With Grade 1 Cystitis, Assessed by CTCAE v3.0, During Concurrent Valproic Acid and Radiation Treatment
Description: document frequency of grade 2 cystitis, assessed by CTCAE v3.0, during concurrent valproic acid and radiation treatment from week 1-10
Time Frame: first 10 weeks of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

18. Primary Outcome: Percentage of Participants With Grade 3 Thrombocytopenia, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 3 thrombocytopenia, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 3

19. Primary Outcome: Percentage of Participants With Grade 3 Neutropenia, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 3 neutropenia, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 3

20. Primary Outcome: Percentage of Participants With Grade 3 Lymphopenia, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 3 lymphopenia, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 3

21. Primary Outcome: Percentage of Participants With Grade 2 Intratumoral/Intracranial Hemorrhage, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 2 intratumoral/intracranial hemorrhage, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

22. Primary Outcome: Percentage of Participants With Grade 3 Fatigue, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: Document frequency of grade 3 fatigue, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 3

23. Primary Outcome: Percentage of Participants With Grade 2 Fatigue, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 2 or higher fatigue, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 7

24. Primary Outcome: Percentage of Participants With Grade 3 Somonolence, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: Document frequency of grade 3 somonolence, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

25. Primary Outcome: Percentage of Participants With Grade 2 Somonolence, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 2 somnolence, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 2

26. Primary Outcome: Percentage of Participants With Grade 3 Weight Gain, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: Document frequency of grade 3 weight gain, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 2

27. Primary Outcome: Percentage of Participants With Grade 2 Weight Gain, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of 2 weight gain, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

28. Primary Outcome: Percentage of Participants With Grade 3 Hypertension, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 3 hypertension, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 4

29. Primary Outcome: Percentage of Grade 2 Hypertension, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: Document frequency of grade 2 hypertension, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 8

30. Primary Outcome: Percentage of Participants With Grade 2 Hypoglycemia, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 2 hypoglycemia, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

31. Primary Outcome: Percentage of Participants With Grade 3 Subacute Bone Infarction, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 3 subacute bone infarction, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

32. Primary Outcome: Percentage of Participants With Grade 3 Cellulitis, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 3 cellulitis, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

33. Primary Outcome: Percentage of Participants With Grade 2 Proteinuria, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 2 proteinuria, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 2

34. Primary Outcome: Percentage of Participants With Grade 4 Deep Vein Thrombosis, Pulmonary Embolism, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 4 deep vein thrombosis, pulmonary embolism, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

35. Primary Outcome: Percentage of Participants With Grade 2 Ocular Keratitis, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 2 ocular keratitis, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

36. Primary Outcome: Percentage Participants With Grade 2 Urinary Tract Infection, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 2 urinary tract infection, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

37. Primary Outcome: Percentage of Participants With Grade 2 Cough, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 2 cough, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

38. Primary Outcome: Percentage of Participants With Grade 2 Anorexia, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 2 anorexia, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 3

39. Primary Outcome: Percentage of Participants With Grade 2 Hypoalbuminemia, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 2 hypoalbuminemia, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 3

40. Primary Outcome: Percentage of Participants With Grade 2 Abdominal Pain, Assessed by CTCAE v3.0, During Maintenance Therapy of Valproic Acid and Bevacizumab
Description: document frequency of grade 2 abdominal pain, assessed by CTCAE v3.0, during maintenance therapy of valproic acid and bevacizumab, from week 11 to up to 24 months
Time Frame: from week 11 to up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | 38 Eligible Patients
Number analyzed (Participants) | 38
Participants | 1

41. Secondary Outcome: Median Event Free Survival (EFS)
Description: estimate the median event free survival of patients receiving protocol therapy
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Diffuse Intrinsic Pontine Glioma | High-grade Gliomas
Number analyzed (Participants) | 19 | 17
months | 7.8 [5.6 to 8.2] | 9.1 [6.4 to 11]
Statistical Analysis 1: Comparison: Diffuse Intrinsic Pontine Glioma; Test type: Other — The Kaplan-Meier method was used to estimate the median EFS for each cohort with 95% confidence intervals. All analyses were performed in SAS version 9.4 statistical software (SAS Institute Inc) and R (https://cran.r-project.org/); The Kaplan-Meier method was used to estimate the median EFS for each cohort with 95% confidence intervals

42. Secondary Outcome: Median Overall Survival (OS)
Description: median OS of patients receiving protocol therapy
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Diffuse Intrinsic Pontine Glioma | High-grade Gliomas
Number analyzed (Participants) | 19 | 17
months | 10.3 [7.4 to 13.4] | 12.1 [10 to 22.1]
Statistical Analysis 1: Comparison: Diffuse Intrinsic Pontine Glioma vs High-grade Gliomas; Test type: Other — The Kaplan-Meier method was used to estimate the one-year EFS for each cohort with 95% confidence intervals. All analyses were performed in SAS version 9.4 statistical software (SAS Institute Inc) and R (https://cran.r-project.org/); The Kaplan-Meier method was used to estimate the one-year EFS for each cohort with 95% confidence intervals

43. Secondary Outcome: Partial Response in Diffuse Intrinsic Pontine Glioma
Description: partial response defined as 51% to 99% reduction in tumor size,determined using WHO bi-dimensional criteria (product of the greatest tumor diameter and its perpendicular diameter)
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Diffuse Intrinsic Pontine Glioma: 20 eligible patients, 16 evaluable patients
Arm/Group | Diffuse Intrinsic Pontine Glioma
Number analyzed (Participants) | 16
Participants | 8
Statistical Analysis 1: Comparison: Diffuse Intrinsic Pontine Glioma; partial response defined as 51% to 99% reduction in tumor size,determined using WHO bi-dimensional criteria (product of the greatest tumor diameter and its perpendicular diameter); Test type: Other; Not applicable (8 partial responses in 16 patients = 50%)

44. Secondary Outcome: Partial Response in High-grade Gliomas
Description: as for outcome 43
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Groups:
- High-grade Gliomas: 18 eligible patients, 14 evaluable patients
Arm/Group | High-grade Gliomas
Number analyzed (Participants) | 14
Participants | 5

45. Secondary Outcome: Complete Response in High-grade Gliomas
Description: complete response defined as complete disappearance of all measurable lesions,determined using WHO bi-dimensional criteria (product of the greatest tumor diameter and its perpendicular diameter)
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | High-grade Gliomas
Number analyzed (Participants) | 14
Participants | 1

ADVERSE EVENTS:
Time Frame: up to 24 months
Arm/Group | 38 Eligible Patients
All-Cause Mortality (participants affected / at risk) | 37/38
Serious Adverse Events (participants affected / at risk) | 4/38
Other Adverse Events (participants affected / at risk) | 33/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 38 Eligible Patients (N=38)
radiation necrosis (Nervous system disorders) | 1 (1) — radiation necrosis during concurrent valproic acid and radiation therapy
amylase and lipase elevation (Gastrointestinal disorders) | 1 (1) — patient had grade 3 amylase and lipase elevation with clinical vomiting/anorexia at week 10 of protocol therapy
subacute bone infarction (Musculoskeletal and connective tissue disorders) | 1 (1) — grade-3 subacute bone infarction and cellulitis while receiving valproic acid and bevacizumab
intratumoral hemorrhage (Nervous system disorders) | 1 (1) — grade-2 (clinically asymptomatic) intratumoral hemorrhage (in a patient with DIPG) while receiving valproic acid and bevacizumab
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 38 Eligible Patients (N=38)
thormbocytopenia (Blood and lymphatic system disorders) | 3 (5) — grade-3 thrombocytopenia
neutropenia (Blood and lymphatic system disorders) | 3 (4) — grade-3 neutropenia
lymphopenia (Blood and lymphatic system disorders) | 3 (3) — grade-3
somnolence (Nervous system disorders) | 3 (4) — 2 grade-2 and 1 grade-3 somnolence
fatigue (Nervous system disorders) | 10 (11) — 7 grade-2 and 3 grade-3 fatigue
weight gain (Metabolism and nutrition disorders) | 3 (5) — 1 grade-2 and 2 grade-3 weight gain
hypertension (Cardiac disorders) | 12 (18) — 8 grade-2 and 4 grade-3 hypertension
proteinuria (Renal and urinary disorders) | 2 (2) — 2 grade-2 proteinuria
anorexia (Metabolism and nutrition disorders) | 3 (3) — 3 grade-2 anorexia
hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) — 3 grade-2 hypoalbuminemia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-09-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT00879437/Prot_SAP_ICF_000.pdf